CLINICAL TRIAL: NCT06429358
Title: The Role of Probiotics in Preventing Recurrent Urinary Tract Infections in Pregnant Women: A Randomized Control Trial
Brief Title: The Role of Probiotics in Preventing Recurrent Urinary Tract Infections in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frontier Medical and Dental College, Abbotabad (Other)
Responsible Party: Principal Investigator, Dr Saif ur Rehman, Professor, Frontier Medical and Dental College, Abbotabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3388
Record Dates: First submitted 2024-05-15; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Experimental): The probiotic group received a daily oral supplement with Lactobacillus rhamnosus. The probiotic supplement was delivered as easy-to-swallow capsules.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus
- Control Group (Other)
  Interventions: Other: Control Group

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus — The probiotic supplement was delivered in the form of easy-to-swallow capsules.
  Arms: Probiotic Group
Other: Control Group — Participants in the control group were given a placebo that looked, tasted, and felt just like the probiotic pill.
  Arms: Control Group

SUMMARY:
Urinary tract infections (UTIs) are a significant public health problem affecting more than 150 million people worldwide and causing a significant economic impact of approximately US$ 6 billion annually. It is one of the most common infectious diseases after upper respiratory tract infections. More than 50% of women and at least 12% of men will be affected by urinary tract infections in their lifetime. The probiotic supplement was delivered as easy-to-swallow capsules specifically prepared to maintain the viability and stability of the Lactobacillus rhamnosus GG strain throughout the research period. Participants were told to take the probiotic supplement with water to maximise absorption and efficiency, ideally after meals.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18-40 year
* History of recurrent urinary tract infections (two or more episodes in the past year).
* Singleton pregnancy.

Exclusion Criteria:

* Multiple gestations.
* History of preterm labor.
* Chronic medical conditions (e.g., diabetes mellitus, immunodeficiency disorders).
* Use of antibiotics or probiotics within the past month.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 14 week's gestation with diagnosed UTI
Enrollment: 30 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Urinary Detailed Report Values | second trimester of pregnancy (about 14 week's gestation) and lasted until birth, a period of roughly 26 to 28 weeks.
  The test was performed to determine levels of neutrophils
Urine Culture | second trimester of pregnancy (about 14 week's gestation) and lasted until birth, a period of roughly 26 to 28 weeks.
  Urine Culture:
  Urine samples were collected aseptically prior to and after intervention and cultured to detect bacterial pathogens linked with urinary tract infections. This assessment was carried out at two distinct time points:
  Pre-Intervention: Before beginning the probiotic intervention, baseline urine samples were taken to detect any existing bacterial illnesses and create a point of comparison.
  Post-Intervention: After the intervention period, individuals supplied an additional urine sample for culture investigation. This post-intervention evaluation sought to establish any changes in the prevalence of bacterial pathogens, particularly those known to cause urinary tract infection
Leukocytes: | second trimester of pregnancy (about 14 week's gestation) and lasted until birth, a period of roughly 26 to 28 weeks.
  leukocytes in urine were evaluated
Nitrites: | second trimester of pregnancy (about 14 week's gestation) and lasted until birth, a period of roughly 26 to 28 weeks.
  presence of nitrites in urine before and after intervention was investigated
pH | second trimester of pregnancy (about 14 week's gestation) and lasted until birth, a period of roughly 26 to 28 weeks.
  Urinary pH values were measured

CONTACTS AND LOCATIONS:
Locations (1):
- Frontier Medical and Dental College, Abbottābād, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No